CLINICAL TRIAL: NCT03047239
Title: A Prospective Study Investigating the Relationship Between SENSIMED Triggerfish® Ocular Dimensional Profiles and Disease Progression in Patients With Open Angle Glaucoma
Brief Title: TF for the Prediction of Visual Field Progression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: strategic change
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1701
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open angle glaucoma (Experimental): SENSIMED Triggerfish
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Smart contact lens based device indicated to detect the peak patterns of variation in intraocular pressure over a maximum period of 24 hours

SUMMARY:
Baseline 24-hour SENSIMED Triggerfish (TF) recordings as well as functional and structural vision tests measured prospectively every 3 months over a 2-year period, will be used to model TF's ability to serve as a risk factor for individual progression rates.

DETAILED DESCRIPTION:
Glaucoma subjects will be selected based on scheduled appointments (consecutive selection) and clinic records such as patient databases (convenience selection) and invited to participate in the study. After having signed and dated the informed consent form, they will receive an appointment for a screening visit, during which they will undergo an ophthalmic examination and review of their medical and ophthalmic history as well as prior and current treatments. The eye at higher risk of disease progression will be selected for the study if both eyes are eligible.

On study day 0 (SD0), subjects will receive TF for a 24-hour recording of the profile of ocular dimensional changes, starting between 11 am and 3 pm, with simultaneous recording of 24-hour blood pressure (BP). The recordings will be carried out in ambulatory conditions with the subjects pursuing as close to normal daily activities as possible. Subject activities will be captured in a logbook. After completion of the recording, subjects will receive an ophthalmic exam to exclude or adequately address any side effects and provide the logbook to the investigator.

At 3-month intervals following the TF recording until 2 years after the TF recording, follow-up visits will be scheduled for assessment of the visual field (VF), the retinal nerve fiber layer (RNFL) thickness by optical coherence tomography (OCT), optic disc photo and intraocular pressure (IOP). 24-hour TF recording (starting at the same time as on SD0) will be performed at 1 and 2 years and, if glaucoma subjects undergo a glaucoma surgery in the follow-up period, an additional 24-hour TF profile will be recorded approximately 3 months after the intervention (again starting at the same time as on SD0).

ELIGIBILITY:
Inclusion Criteria:

1. For glaucoma subjects, a clinical diagnosis of OAG* in the study eye with an abnormal optic disc defined as:

   * diffuse or focal narrowing, or notching, of the optic disc rim, or
   * progressive narrowing of the neuroretinal rim with an associated increase in cupping of the optic disc increased cupping of the optic disc, or
   * diffuse or localized abnormalities of the parapapillary RNFL, or
   * disc rim, parapapillary RNFL, or lamina cribrosa hemorrhages, or
   * optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue, or
   * large extent of parapapillary atrophy and an abnormal VF defined as
   * VF damage consistent with RNFL damage (e.g., nasal step, arcuate field defect, or paracentral depression in clusters of test sites) based on the presence of a cluster of 3 or more non-edge points on the pattern deviation plot at p < 5% with 1 point at p < 1%, or
   * Glaucoma Hemifield Test (GHT) outside normal limits.

     * OAG*:

       * Primary open angle glaucoma (POAG; includes normal tension glaucoma (NTG), i.e.: POAG with all known untreated IOP measurements < 22 mmHg using Goldmann applanation tonometry): defined by the presence of open angles on gonioscopy in the absence of other causes of glaucomatous optic neuropathy and VF defects; or
       * Exfoliative glaucoma (XFG): defined by the presence of exfoliative material on the pupil border and/or on the surface of the lens capsule except the central zone; or
       * Pigmentary glaucoma (PEG): defined by the presence of pigment dispersed on the trabecular meshwork, Schwalbe's line, the iris surface, the lens equator, the corneal endothelium, and/or characteristic trans-illumination defects of the mid-peripheral iris.
2. For glaucoma subjects, MD not worse than -12.00 dB at enrollment in the study eye
3. For glaucoma subjects, no IOP-lowering treatment or stable IOP-lowering treatment regimen in the study eye in the 3 months prior to the screening visit
4. For glaucoma subjects, at least 1 year of experience with VF testing
5. For healthy subjects, normal optic disc, normal VF, IOP ≤ 21 mmHg and open anterior chamber angle in the study eye and no known family history of glaucoma
6. Best corrected visual acuity (BCVA) 20/25 in the study eye at time of screening
7. Aged 22 to 80 years
8. Spherical and cylinder equivalent in the study eye between ±6.00 and ±3.00 diopters, respectively
9. Having given written informed consent, prior to any investigational procedures

Exclusion Criteria:

1. Ocular pathology other than glaucoma in the study eye affecting VF test and OCT-RNFL results
2. Glaucoma surgery in the study eye prior to the screening visit
3. Cataract surgery or glaucoma laser treatment in the study eye within 3 months of the screening visit
4. Subjects with allergy to corneal anesthetic
5. Subjects with contraindications for TF wear: active eye disease, eye injury or eye abnormality affecting the cornea, conjunctiva, or eyelids, subject history of eye or eyelid infections including styes or history of AEs associated with wearing contact lenses, or intolerance, or abnormal ocular response to contact lenses, active inflammation of the eye, active infection of the eye, corneal vascularization, insufficiency of lacrimal secretion, corneal hypoesthesia, known allergy to silicone
6. Subjects unable or unwilling to comply with the study procedures and who are unlikely to be able to complete the 24-month follow-up period.
7. Participation in other interventional clinical research within the last 4 weeks

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic odds ratio (DOR) for a SENSIMED Triggerfish based model for the prediction of visual field annual progression rate (24-2 SITA Standard) measured as Mean Deviation (MD) slope | 2 years

IPD SHARING:
Plan to Share IPD: No